CLINICAL TRIAL: NCT04533178
Title: Posterior Lumbar Stress Reaction in Pediatric Patients. Treatment With or Without Soft Spinal Brace?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Kari Kangassalo, Principal investigator, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T102/2020
Record Dates: First submitted 2020-04-16; First posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Back Pain; Stress Fracture
Keywords: stress reaction; spinal brace
MeSH Terms: conditions — Back Pain; Fractures, Stress

STUDY DESIGN:
Intervention Model Description: Multicenter study comparing treatment with or without soft spinal brace
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restriction of sports activities (Active Comparator): No sports during the 6 week treatment period
  Interventions: Other: Resting from all sports activities
- Restriction of sports activities and soft spinal brace (Experimental): No sports and use of a soft spinal brace 16 hours per day during the 6 week treatment period
  Interventions: Device: soft spinal brace; Other: Resting from all sports activities

INTERVENTIONS:
Device: soft spinal brace — Use of a soft spinal brace 16 hours per day during the 6 week treatment period.
  Arms: Restriction of sports activities and soft spinal brace
Other: Resting from all sports activities — Resting from all sports activities

SUMMARY:
A clinical trial will be conducted comparing healing of a posterior lumbar vertebra stress reaction in children treated either with cessation of sports activities for a period of six weeks and wearing a soft spinal brace 16 hours per day or cessation of sports activities only. Primary outcome is the change in stress reaction on MRI at 6 weeks compared to pre-treatment MRI.

DETAILED DESCRIPTION:
A clinical trial will be conducted comparing healing of an acute posterior lumbar vertebra stress reaction in children treated either with cessation of sports activities for a period of six weeks and wearing a soft spinal brace 16 hours per day or cessation of sports activities only. Inclusion criteria will be a child or an adolescent aged between 8 and 18 years with a posterior lumbar vertebra stress reaction uni- or bilaterally in one or more lumbar vertebra. Bone marrow edema in the dorsal parts of the lumbar spine must be confirmed in a recent (under 3 weeks) MRI examination. Exclusion criteria will be a fracture line (spondylolysis), spondylolisthesis or other abnormalities on lumbar CT examination. Other exclusion criteria are skeletal disorder or not consenting to be a patient in this study.

110 Patients/ participants are randomized into two groups. The first group of 55 patients is treated with cessation of all sports activities and a soft spinal brace. The other group is treated only with cessation of sports activities. Treatment in both groups is 6 weeks, starting at doctor's appointment after all necessary examinations are complete. Minimum follow-up will be 6 months.

In the beginning of this study a blood plasma vitamin D values will be measured from all our patients. Patients with D-vitamin values below 50 nmol/l will receive vitamin D prescription.

Lateral x-ray picture of the lumbar spine is taken with axial loading (standing) from all study patients at the beginning and at the end (6 months) of the study. This enables to see the possible change in sacral slope during the 6-month follow-up. The possible change will then indicate a change in lumbar posture during this time. This is important to clarify whether lumbar posture has a role in the etiology - and treatment - of lumbar vertebra stress injury.

According to statistical power analysis a total of 110 patients - 55 in each group- will be needed to provide evidence for the effectiveness or no effectiveness of a soft spinal brace on the natural history of pars interarticularis stress reaction.

Primary outcome is the change in stress reaction on MRI at 6 weeks compared to pre-treatment MRI.

Secondary outcomes are:

1. SRS-24 - (Scoliosis Research Society) score at the beginning of the treatment and during the six-month follow-up ( at 0, 6 weeks, 6 months appointments)
2. Back and lower extremity pain at the beginning of the treatment and during the six months follow-up (pain drawing including VAS-score (Visual Analogue Pain Score) in children under 16 years old, Oswestry disability index including VAS-score in patients over 16 years old)
3. Relapse of symptoms during the six months follow-up
4. Vitamin D values at the beginning of the study
5. "Pain time table" during the 6-week period of treatment - to clarify the moment of ending of pain during treatment.
6. Change in sacral slope on lateral lumbar x-ray with axial loading during the 6 months of follow-up.
7. Pain in one-legged back extension test at 0, 6 weeks and 6 months follow-up appointments

ELIGIBILITY:
Inclusion Criteria:

* Uni- or bilateral acute stress reaction of pars interarticularis or other part of posterior lumbar vertebra on MRI
* No signs of fracture line on MRI or CT
* Age between 8 and 18 years
* Written informed consent
* Low back pain

Exclusion Criteria:

* Spondylolysis
* Spondylolisthesis
* Systemic skeletal disorder (Osteogenesis imperfecta, skeletal dysplasia), osteoporosis
* Systemic diseases (e.g. Diabetes mellitus type 1, rheumatic diseases, inflammatory bowel diseases, Marfan syndrome)
* Other bony abnormalities seen on lumbar MRI examination (e.g. Scheuermann disease, L5 sacralisation, spina bifida)

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in stress reaction | 6 weeks
  Change in stress reaction on MRI at 6 weeks compared to pre-treatment MRI

SECONDARY OUTCOMES:
SRS-24 -score at the beginning of the treatment and during the six-month follow-up | 6 months
  Change in SRS-24 (Scoliosis Research Society patient outcome) questionnaire score during the six month follow-up; Total amount of points possible from each visit questionnaire is 120, divided by the number of questions (max 24, depending on number of questions answered). This results in the final score that can vary from 1 to 5, where 5 is the best and 1 is the worst.
Back pain | six months
  Pain drawing in children under 16 years, Oswestry disability index in children over 16 years.
Relapse of symptoms | six months
  Relapse of symptoms during the six month follow-up
Vitamin D value | Only at start of study. The blood test for Vitamin D is taken at the first appointment / day of recruitment to this study, which is day 1 of the study.
  Vitamin D value (D25 Hydroxy test) is measured at the time of the first study visit, at baseline. A value below 30 ng/ml is considered low. If the value is below 30 ng/mol, total Vitamin D supplement (20 mcg/day) is prescribed for a minimum of 3 months. This is to ensure adequate Vitamin D levels for all study subjects required for bone fracture healing.
Duration of pain during treatment | six weeks
  "pain time table" filled by the patient during the 6 week treatment period
change in sacral slope | six months
  Change in sacral slope on lateral lumbar x-ray with axial loading during the 6 months of follow-up
pain in one-legged back extension test | six months
  pain in one-legged back extension test at 0, 6 week and 6 month follow-up appointments

CONTACTS AND LOCATIONS:
Locations (4):
- Finland (4):
  - Tampere University Hospital, Tampere, Pirkanmaa
  - SataSairaala, Pori, Satakunta
  - Turku University Hospital, Turku, Southwest Finland
  - Mehilainen Neo Turku, Turku, Southwest Finland

IPD SHARING:
Plan to Share IPD: No
Not necessary